CLINICAL TRIAL: NCT03042650
Title: Intensive Referral to Reduce Smoking in Probationers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0018-16-FB
Record Dates: First submitted 2016-12-29; First posted 2017-02-03 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Smoking Cessation; Substance Use Disorder
MeSH Terms: conditions — Smoking Cessation; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Referral Intervention Group (Experimental): Intensive Referral Intervention will by done by trained probation officers
  Interventions: Behavioral: Intensive Referral Intervention Group
- Standard Practice Facilitated Group (Active Comparator): Standard Current Practice will be provided by untrained probation officers
  Interventions: Behavioral: Standard Practice Facilitated Group

INTERVENTIONS:
Behavioral: Intensive Referral Intervention Group — The Intensive Referral Intervention Group will review a series of pamphlets regarding participation in 12-step meetings as well as smoking cessation that will be presented in a group setting to probationers in 3 sessions.
  Arms: Intensive Referral Intervention Group
Behavioral: Standard Practice Facilitated Group — The Standard Practice Facilitated Group will receive 3 sessions of the current standard practice for facilitated groups.
  Arms: Standard Practice Facilitated Group

SUMMARY:
The purpose of this study is to determine if Intensive Referral Intervention increases motivation to quit cigarette smoking and quitting-related behaviors in probationers and also to determine if Intensive Referral Intervention improves short-term substance use outcomes in probationers with substance use disorder.

DETAILED DESCRIPTION:
This is a longitudinal study of adults on probation who have a Substance Use Disorder (SUD) and smoke cigarettes. One-half of probation officers will be trained in the Intensive Referral Intervention (IRI) while one-half will deliver Standard Practice which is to encourage support group attendance. Research staff will assess fidelity to the IRI in trained probation officers. The investigators propose to enroll 150 probationers over a four month period and complete 3 and 6-month follow-up interviews to assess smoking and substance use measures.

ELIGIBILITY:
Inclusion Criteria:

* CBR-MH Probationers in Douglas County, NE
* SUD
* daily cigarette smoker

Exclusion Criteria:

* Under guardianship
* unwilling to provide personal contact information
* unable to pass Mini-Cog

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Motivation measured by Fagerstrom Test | 6 Months
  Increased Motivation to quit cigarette smoking in probationers as indicated by change in Fagerstrom Test for Nicotine Dependence

SECONDARY OUTCOMES:
Change in Timeline Follow-back Calendar | 6 Months
  Improved short term substance use outcomes as indicated by change in Timeline Follow-back Calendar

OTHER OUTCOMES:
Motivation measured by Readiness to Quit Ladder | 6 Months
  Increased Motivation to quit cigarette smoking in probationers as indicated by a change in Readiness to Quit Ladder
Motivation measured by QSU-Brief Questionnaire for Smoking Urges | 6 Months
  Increased Motivation to quit cigarette smoking in probationers as indicated by a change in QSU-Brief Questionnaire for Smoking Urges

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Grant, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No